CLINICAL TRIAL: NCT04617353
Title: Experience With the Combined Method of Air-plasma Flow and Nitric Oxide Therapy in the Prevention and Treatment of Wound Infectious Complications in Cardiac Surgery
Brief Title: Combined Air-plasma Flow and Nitric Oxide Therapy in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TomskNRMC
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Mediastinitis
Keywords: plasma; endogenous nitric oxide; infectious complications; mediastinitis
MeSH Terms: conditions — Mediastinitis

STUDY DESIGN:
Intervention Model Description: Patient enrollment according to the inclusion criteria. Carrying out medical manipulations according to the group inclusion criteria. Efficiency control based on the clinical course of the disease, instrumental and laboratory study methods.
  After the patient is discharged from the hospital, a follow-up examination after 12 months, including an objective examination, a spiral computed tomography of the chest organs. Complete blood count, general urine test, biochemistry blood test.
  Comparison of the main clinical and laboratory parameters between patients of both groups: the total number of bed-days spent, the time spent in the ICU, the duration of mechanical ventilation, laboratory parameters: red blood cell count, coagulation system, markers of infection and inflammation, state of sepsis, determination of how fast the bone tissue reparation is. CT scan of the chest, sternum, examination of the bacterial flora and bacterial contamination of the postoperative wound
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma (Experimental): (the treatment of sterno-mediastinitis was carried out using a combined method of air-plasma flow and NO therapy)
  Interventions: Procedure: NO-based treatment of sterno-mediastinitis
- Standard therapy (Other): (patients who were treated for sterno-mediastinitis according to clinical guidelines, the main method of which is a permanent irrigation and aspiration flow drainage method, as well as a Vacuum Assisted Closure (VAC) system of dressings for vacuum drainage)
  Interventions: Procedure: Treatment of sterno-mediastinitis

INTERVENTIONS:
Procedure: NO-based treatment of sterno-mediastinitis — Preparation of a postoperative wound in case of infectious complications. A mandatory sampling material for culture and antibiotic sensitivity is collected before and after the air plasma flow treatment.
  Direct effect of the air-plasma flow on the entire wound surface in sterilization mode with an exposure of 2-3 minutes for each surgical wound, until the level of bacterial contamination decreases to 10-5 and below.
  The technique of using air-plasma flow when closing a wound after preventing infectious complications in it.
  In the postoperative period, daily air-plasma flow treatment in sterilization mode along the suture line for 3 minutes. Penetrating drainage NO supply in the biological stimulation mode daily for 10 days, with an exposure of 1-2 minutes up to 10 days, with a volume of up to 2 liters per minute.
  Collecting wound culture from the drainage containers on 1-3-7-12 days to detect pathogens and the bacterial number.
  Arms: Plasma
Procedure: Treatment of sterno-mediastinitis — patients who were treated for sterno-mediastinitis according to clinical guidelines, the main method of which is a permanent irrigation and aspiration flow drainage method, as well as a Vacuum Assisted Closure (VAC) system of dressings for vacuum drainage
  Arms: Standard therapy

SUMMARY:
In cardiovascular surgery, the most common and serious complication is postoperative wound infection. The most formidable wound complication is mediastinitis, the frequency of which varies from 1 to 3%. Currently, mortality in this group of patients varies from 3.5 to 58.3%. In this regard, the relevance of developing new methods for the prevention and treatment of infectious wound complications is beyond doubt. In this study, it is supposed to examine and evaluate the effectiveness of the combined effects of air-plasma flow and nitric oxide in the treatment of postoperative infectious complications in cardiac surgery.

DETAILED DESCRIPTION:
One of the most common and serious complications in cardiovascular surgery is sternal wound infection. According to many authors, the incidence of infectious complications after sternotomy ranges from 0.4% to 15% . Superficial infection of the anterior chest wall after median sternotomy occurs in 0.4-15% . Typically, this complication is detected within the first two weeks (on average, about seven days). The most formidable wound infectious complication is mediastinitis. According to various authors, the incidence of mediastinitis varies from 1 to 3%. Mortality in this group of patients reaches 39% . Until now, the only effective and generally accepted method for treating patients with mediastinitis has been antibiotic therapy in combination with surgical intervention. The options for antibiotic therapy remain generally accepted and their effectiveness is not discussed, however, there are many options for various types of surgical treatment. Their main principle is to perform resternotomy, necrosectomy, followed by reosteosynthesis of the sternum and the installation of permanent irrigation and aspiration, flow-through drainage. Despite this, the mortality rate in this pathology remains invariably high. In this regard, issues related to the development of new medical technologies, methods for prevention and treatment of infectious wound complications do not lose their relevance at the present time.

During the study, it is supposed to use an original method developed for the prevention, as well as for the treatment of wound infectious complications.

The advantage of the investigator's proposed original method of treating mediastinitis is in the combined effect of thermal (air-plasma flow) and biochemical (effect of NO on wound surfaces) by stimulating the processes of regeneration and repair.

Also, for obvious reasons, resistance cannot arise to it, which is relevant in the context of the widespread transmission of nosocomial infections, especially in large hospitals, such as modern cardiology dispensaries.

As a result of the work, the cases of infectious wound complications in the early postoperative period, the total number of bed-days spent, the time spent in the ICU, the duration of mechanical ventilation, laboratory parameters: red blood cell count, coagulation system, markers of infection and inflammation, state of sepsis, determination of how fast the bone tissue reparation is, CT scan of the chest, sternum, examination of the bacterial flora and bacterial contamination of the postoperative wound will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent heart and great vessels surgery with confirmed laboratory, bacteriological, instrumental tests, as well as the presence of clinical signs of sterno-mediastinitis.
* Signed informed consent to participate in the study

Exclusion Criteria:

* Patients who underwent heart and great vessels surgery not through a median sternotomy.
* Patients who have signs of inconsistency of sutures or any other wound complications, but there are no clinical, laboratory, bacteriological data indicating infection of the postoperative wound.
* No informed consent to participate in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Death | 30 days
  In-hospital mortality rate (%)
Re-infection of the wound | 30 days
  Rate wound re-infection (%)
Skin suture incompetence | 30 days
  Rate of skin suture incompetence (%) due to lack of tissue repair
Recovery | 30 days
  Rate of full recovery (%)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kuznetsov, PhD, Study Chair — Tomsk National Research Medical Center of the Russian Academy of Sciences
Locations (1):
- TomskNRMC, Tomsk, Tomskay Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.